CLINICAL TRIAL: NCT02930239
Title: Early Initiated Gait Rehabilitation Using the Anti-gravity Treadmill Following an Anterior Cruciate Ligament Reconstruction
Brief Title: Gait Rehabilitation Following an Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Joanna Kvist, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dnr 2016/25-31
Record Dates: First submitted 2016-02-08; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Complete Tear, Knee, Anterior Cruciate Ligament
Keywords: ACL-reconstruction; Gait rehabilitation; Anti Gravity treadmill; ACL-rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gait rehabilitation (Experimental): Will perform 2 weeks of gait rehabilitation using the anti gravity treadmill. Intervention will start 2 weeks post-surgery. This rehabilitation will be performed simultaneously as the patient receives the standardized rehabilitation at Linkoping University Hospital.
  Interventions: Other: Gait rehabilitating with reduced bodyweight; Other: Standardized rehabilitation following an anterior cruciate ligament reconstruction at Linkoping University Hospital
- Control group (Active Comparator): Will only receive the standardized rehabilitation at Linkoping University Hospital.
  Interventions: Other: Standardized rehabilitation following an anterior cruciate ligament reconstruction at Linkoping University Hospital

INTERVENTIONS:
Other: Gait rehabilitating with reduced bodyweight — Patients will perform 8 sessions of gait rehabilitation with reduced bodyweight using the anti gravity treadmill during week 2-5 post-surgery.
  Arms: Gait rehabilitation
Other: Standardized rehabilitation following an anterior cruciate ligament reconstruction at Linkoping University Hospital — Exercises for increased movement and circulation performed on a daily basis.

SUMMARY:
A randomized control trial where subjects following an anterior cruciate ligament reconstruction will be randomized to either a control group who will receive the normal rehabilitation or an experimental group who will perform a 2-week gait rehabilitation using the anti-gravity treadmill in addition to the normal rehabilitation. The intervention will be added to the existing care received at Linkoping University Hospital 2 weeks post-surgery, while the evaluation will be performed in week 5 and 12 post-surgery using: a 3D-gait analysis (with the Qualisys software), self-reported function questionnaires and a clinical examination.

ELIGIBILITY:
Inclusion Criteria:

* Anterior cruciate ligament injury occurred a minimum of 3 weeks prior to surgery

Exclusion Criteria:

* Previous Anterior cruciate ligament injury
* Other knee injury with restrictions that could interfere with rehabilitation
* Other injury or disease that could interfere with rehabilitation
* Inability to understand the information

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-07 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
3 dimensional gait analysis | 5 weeks post-surgery
  A 10 Oqus camera system by Qualisys, Sweden integrated with 3 Kistler forcplates is used. The primary outcome is peak knee flexion during stance phase for injured leg

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | 5 weeks post-surgery
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is a self-administered questionnaire which consists of 42 items which can be sub grouped into five categories. These categories are pain, other disease-specific symptoms, activities of daily living (ADL), sport and recreation function and lastly knee-related quality of life.
International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) | 12 weeks post-surgery
  The IKDC subjective knee evaluation form is a self-administered questionnaire which contains 18 items divided into 3 subgroups. These subgroups are symptoms, sports and daily activities and the patients current and previous levels of knee function.
3 dimensional gait analysis | 12 weeks post-surgery
  A 10 Oqus camera system by Qualisys, Sweden integrated with 3 Kistler forcplates is used. The primary outcome is peak knee flexion during stance phase for injured leg

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kvist, Professor, Principal Investigator — Linkoeping University
Locations (1):
- Linkoping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No